CLINICAL TRIAL: NCT07320885
Title: Fiber-Reinforced Versus Bulk-Fill Flowable Resin Composite Dentin Replacement Materials: 4-Year Clinical Performance in Class II Cavities
Brief Title: Clinical Performance of Fiber-Reinforced Dentin Replacement Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Youness Saleh, lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A11120520
Record Dates: First submitted 2025-11-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Caries; Dentin; Caries Class II
Keywords: Fiber-reinforced resin composite; Flowable bulk-fill resin composite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ever x flow short-fiber reinforced composite (Experimental): Ever x flow was used as dentin replacement material in class II cavities
  Interventions: Other: Ever x flow
- SDR flowable bulk-fill resin composite (Experimental): SDR was used as dentin replacement material
  Interventions: Other: SDR
- Tetric N-Flow Bulk fill resin composite (Experimental): Tetric N-Flow Bulk fill was used as dentin replacement material
  Interventions: Other: Tetric N-Flow Bulk fill

INTERVENTIONS:
Other: Ever x flow — Ever x flow was used as dentin replacement material
  Other Names: flowable FRC
  Arms: Ever x flow short-fiber reinforced composite
Other: SDR — SDR was used as dentin replacement material in class II cavities
  Arms: SDR flowable bulk-fill resin composite
Other: Tetric N-Flow Bulk fill — Tetric N-Flow Bulk fill was used as dentin replacement material in class II cavities
  Arms: Tetric N-Flow Bulk fill resin composite

SUMMARY:
the current study was conducted to evaluate and compare the flowable short fiber-reinforced (SFRC) and flowable bulk-fill resin composites (BFCs) regarding their 4-year clinical performance as dentin replacement materials in class II cavities.

DETAILED DESCRIPTION:
the current study was conducted to evaluate and compare the flowable short fiber-reinforced (SFRC) and flowable bulk-fill resin composites (BFCs) regarding their 4-year clinical performance as dentin replacement materials in class II cavities. Forty patients were enrolled in the study. Each patient received three class II cavities; one of them was restored with flowable SFRC for dentin replacement, while in the other two cavities, dentin was replaced with two different flowable BFCs. The three dentin replacements were veneered with one particulate filler resin composite (PFC) (Essentia, GC). World Dental Federation (FDI) criteria were used for clinical assessment of the restorations at 1-week (baseline), 6, 12, 18-months, 2, 3, and 4-year intervals.

ELIGIBILITY:
Inclusion Criteria:

* having good oral hygiene.
* having at least 3 posterior teeth with moderate to large primary proximal carious lesions (score 4 or 5 ICDAS).
* ranging in age from 20 to 40 years.
* with normal occlusion.
* accepting to participate in the study by signing an Arabic-written consent according to the regulations of the Mansoura University Ethical Committee.

Exclusion Criteria:

* bad oral hygiene.
* severe chronic periodontitis.
* having installed orthodontic appliances.
* abnormal occlusion.
* parafunctional habits or allergic reaction to any of the materials used in the study.
* teeth with irreversible pulpitis or non-vital teeth.
* fractured or cracked teeth. previously restored teeth.
* teeth with deep sub-gingival cavity margins.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Fracture of restorative material and restoration retention | four years
  Clinical evaluation was performed one week after finishing and polishing (baseline), after 6 months, 1, 2, 3, 4 years using the World Dental Federation (FDI) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
no specific reason